CLINICAL TRIAL: NCT03933254
Title: Intraocular Pressure and Optic Nerve Sheath Diameter Changes in Laparoscopic Cholecystectomies
Status: Withdrawn | Type: Observational
Why Stopped: As a result of COVID-19 pandemics
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assist. Prof., Marmara University
Other Study IDs: 09.2019.264
Record Dates: First submitted 2019-04-27; First posted 2019-05-01 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Intraocular Pressure; Intracranial Pressure; Pneumoperitoneum
Keywords: Intraocular pressure; Optic nerve sheath diameter; Pneumoperitoneum; Laparoscopy; Laparoscopic surgery
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Intraocular pressure measurement via ocular tonometry — Intraocular pressure and optic nerve sheath diameter changes of the patients undergoing laparoscopic cholecystectomy will be measured throughout the surgery at different times using ocular tonometry and ultrasound, respectively.
  Other Names: Optic nerve sheath diameter measurement via ultrasound

SUMMARY:
Pneumoperitoneum created during laparoscopic surgeries has some effects on human physiology. Increased intraabdominal pressure results in increased intrathoracic pressure, and eventually may result in increased intracranial and intraocular pressures. In this study we aimed to identify intraocular and intracranial pressure changes during the perioperative period due to the pneumoperitoneum created for laparoscopic cholecystectomy surgeries. Intraocular pressure will be measured directly from the eye. Intracranial pressure will be estimated by measuring optic nerve sheath diameter changes ultrasonographically.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy
* American Society of Anesthesiologists (ASA) 1 or 2 physical status patients
* Elective surgeries

Exclusion Criteria:

* Patients with glaucoma
* ASA 3 or above patients
* Emergency surgeries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be ASA 1 or 2 physical status patients undergoing elective laparoscopic cholecystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | Throughout the operation (usually about 1 hour).
  The normal physiological value for intraocular pressure is 10-20 mm Hg. It is affected by pneumoperitoneum created for laparoscopy. The pressure will be measured via ocular tonometry through the eye during the surgery at predetermined time intervals.

SECONDARY OUTCOMES:
Intracranial pressure | Throughout the operation (usually about 1 hour).
  The normal physiological value for intracranial pressure is below 10 mm Hg. It is affected by pneumoperitoneum created for laparoscopy. The pressure will be estimated through changes in the optic nerve sheath diameter which will be measured by ultrasonography through the eye during the surgery at predetermined time intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Principal Investigator — Marmara University School of Medicine, Dep of Anesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: No